CLINICAL TRIAL: NCT07003438
Title: Study on the Efficacy and Safety of Fecal Microbiota Transplantation in the Treatment of Steroid - Dependent /Steroid-resistant Nephrotic Syndrome in Children
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhang Ting (Other)
Responsible Party: Sponsor-Investigator, Zhang Ting, chief physician, Shanghai Children's Hospital
Organization: Shanghai Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shanghai Children's Hospital
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Steroid-Resistant Nephrotic Syndrome; Steroid-Dependent Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SDNS:control group (No Intervention): Traditional treatment plan: Steroid Tapering Therapy
- SDNS:Fecal microbiota transplantation group (Experimental): Fecal microbiota transplantation and traditional treatment plan
  Interventions: Drug: Fecal microbiota transplantation (FMT)
- SRNS control group (No Intervention): Conventional treatment plan: Steroid + calcineurin inhibitors (cyclosporine or tacrolimus)
- SRNS:Fecal microbiota transplantation group (Experimental): Conventional treatment plan + fecal microbiota transplantation
  Interventions: Drug: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Drug: Fecal microbiota transplantation (FMT) — FMT was slowly administered to the patient's small intestine with fecal suspension under anesthesia and patients received a second transplant through oral administration freeze-dried capsules containing the fecal matter.
  Other Names: FMT
  Arms: SDNS:Fecal microbiota transplantation group; SRNS:Fecal microbiota transplantation group

SUMMARY:
The objective of this clinical trial was to understand whether FMT is effective in treating steroid-dependent/steroid-resistant nephrotic syndrome in children. It will also learn about the safety of FMT. The main question it was designed to answer was: Did FMT reduce participants '24-hour urine protein content? What medical problems did participants experience while using FMT? The researchers will compare FMT treatment with and without FMT on top of conventional treatment to see if FMT is effective in treating steroid-dependent/steroid-resistant nephrotic syndrome in children. Participants will receive 2 FMT treatments, 1 endoscopic injection under anesthesia, 1 oral fecal bacteria transplantation capsule intake, and follow-up visits (weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48) every 4 weeks from the beginning of medication to our renal specialist clinic for drug efficacy evaluation and safety testing. Blood and fecal samples were collected to determine the effects of fecal bacterial transplantation on intestinal flora, fecal metabolomics, and intestinal mucosal permeability.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-18 years, steroid-dependent/steroid-resistant nephrotic syndrome, regardless of gender, with SDNS at steroid-dependent doses less than 0.5 mg/kg.d

Exclusion Criteria:

* Those with concurrent infections or diseases of other organ systems, and those with abnormal renal function.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
24h urinary protein | follow-up visits (weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48) every 4 weeks from the beginning of medication to our renal specialist clinic for drug efficacy evaluation and safety testing
  24-hour urine protein by urine collection
Gut microbiota | immediately Before FMT, immediately before second FMT, one month after second FMT
  Collect fecal samples
Zonulin | immediately Before FMT, immediately before second FMT, one month after second FMT
  collect blood samples

SECONDARY OUTCOMES:
Serum creatinine | immediately Before FMT, immediately before second FMT, one month after second FMT
  collect blood samples